CLINICAL TRIAL: NCT03451760
Title: Feru-guard (Ferulic Acid and Angelica Archangelica Extract) for Behavioral Symptoms in Dementia
Brief Title: Feru-guard for Behavioral Symptoms in Dementia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Glovia Co., Ltd. (Industry)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17966
Record Dates: First submitted 2018-02-14; First posted 2018-03-02 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Behavioral and Psychiatric Symptoms of Dementia
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled clinical trial with a 12 week intervention period.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind, placebo-controlled study. The placebos will be matched to the active supplement in both sensory and physical characteristics. The participants, study investigators, research associates, and study coordinators will have no knowledge of study assignment. Data analysis will be performed blinded to treatment status. The OHSU Research Pharmacy will be responsible for establishing a randomization scheme for newly enrolled participants. Additionally, the Research Pharmacy will ensure blinding of all study medications. The investigators will also evaluate the effectiveness of our blinding by giving study evaluators, participants, study partners, and investigators a short questionnaire asking about knowledge of group assignment. The randomization code will be broken only after data analysis or if there are numerous serious adverse events before the end of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Feru-guard (Experimental): Over a 12 week period participants will take two 280 mg hard gel capsules of Feru-guard 100M per day (1 capsule am, 1 capsule pm). One capsule will be taken in the morning with a meal and one capsule will be taken in the afternoon with a meal. Each capsule contains 180.32 mg ferulic acid and 20.02 mg of Angelica archangelica. Total daily dose will be 560mg of Feru-guard 100M, with 360.64 mg of ferulic acid and 40.04 mg of Angelica archangelica.
  Interventions: Drug: Feru-guard 100M
- Placebo (Placebo Comparator): Over a 12 week period participants will take two 280 mg hard gel capsules of a placebo per day (1 capsule am, 1 capsule pm). One capsule will be taken in the morning with a meal and one capsule will be taken in the afternoon with a meal.Total daily dosage will be 560mg of a maltodextrin, calcium stearate, and vanilla food flavor mixture.
  Interventions: Other: Feru-guard 100M Placebo

INTERVENTIONS:
Drug: Feru-guard 100M — Feru-guard is a dietary supplement commercially available in Japan in the form of a 1.5 g instant powder packet that is sold in health clinics and directly by Glovia Co. Ltd to patients on doctor's recommendation. The current study will use Feru-guard in the form of a 280 mg hard gel capsule that contains the same amount of the active ingredients (ferulic acid and Angelica archangelica) as the 1.5 g packets. In order to conduct a double-blind, placebo-controlled trial, Feru-guard is contained in opaque, hard gel capsules which allows for better matching of characteristics and improved blinding than studies using powder. Feru-guard will be supplied by Glovia, Co. Ltd., in Tokyo, Japan.
  Arms: Feru-guard
Other: Feru-guard 100M Placebo — In order to conduct a double-blind, controlled trial, the placebo will be contained in opaque, hard gel capsules which allows for better matching of characteristics and improved blinding. The placebo study drug will be matched to the Feru-guard 100M in terms of appearance, smell, and taste.
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
This is designed as a randomized, double-blind, placebo-controlled clinical trial with a 12 week intervention period. Seventy participants with a diagnosis of AD, vascular, and mixed dementia with at least 3 behavioral symptoms present from the Neuropsychiatric Inventory Questionnaires (NPI-Q) will be randomized to the Feru-guard (ferulic acid and Angelica archangelica) or placebo group. Participants will be screened first by a telephone interview or briefly in-clinic and then will be scheduled for an in-clinic screen to establish study eligibility prior to the baseline assessment visit. Clinical and biological outcome measures will occur at baseline and 12 weeks.

DETAILED DESCRIPTION:
The participants will be assessed for eligibility using the NPI-Q and must have at least 3 symptoms present, and a score of 25 or lower on the Mini Mental State Exam (MMSE). Participants will also be screened for a previous diagnosis of either Vascular Dementia, Alzheimer's disease, or Mixed Dementia using DSM-5 criteria. The primary outcome measure will be a change in the total score of Neuropsychiatric Inventory Questionnaire (NPI-Q) over 12-weeks. The investigators expect the group receiving Feru-guard will have a greater improvement in total NPI score compared to the placebo group at 12-weeks.

The investigators will also collect data on the effect of Feru-guard supplementation on care-giver burden using the NPI-Q subscale of caregiver distress, Zarit Burden Interview (ZBI) screening version, and quality of life (SF-12) over 12 weeks. The investigators will also collect data on changes in global cognition of participants over 12 weeks using the Montreal Cognitive Assessment (MoCA). The investigators will compare secondary outcomes between Feru-guard and control group.

ELIGIBILITY:
Inclusion Criteria:

* 55 years old or older.
* Diagnosis of AD, vascular, and mixed dementia
* Neuropsychiatric Inventory Questionnaire (NPI-Q) at least 3 items out of 12 items are rated as "present."
* Use of cholinesterase inhibitors, antidepressants and or antipsychotics medications is allowed, if on stable dosage for at least 2 months.
* Use of memantine and/or serotonin reuptake inhibitors is also allowed, if on stable dose for at least 2 months.
* Have a committed caregiver who is able and willing to assist them with medications, provide study participant information, and attend all study visits.
* Sufficient English language skills to complete all testing.
* MMSE score of 25 or lower.

Exclusion Criteria:

* Participants who started using antipsychotics or anticholinergics within the previous 2 months.
* Participants on blood thinners such as warfarin (Coumadin, jantoven), rivaroxaban (xarelto), fondaparinux (arixtra), dibigatran (pradaxa), apixaban (eliquis) dalteparin (fragmin), enoxaparin (lovenox). Aspirin use is allowed.
* Participants without an identified caregiver.
* Participants with delirium caused by medicinal poisoning or drug intoxication.
* Participants who have had the following diseases before the onset of cognitive impairment:

  1. Alcoholism
  2. Manic depression or bipolar disorder
  3. Schizophrenia
* Participants with malignancy or an acute inflammatory disease.
* Participants with critical circulatory, respiratory, kidney, or liver disease or diabetes.
* BMI of >30.
* Participants who have taken Feru-guard, ferulic acid, or Angelica archangelica supplementation within the last year.
* Enrollment in another clinical trial or treatment study within the previous 6 months.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Neuropsychiatric Inventory Questionnaire at 12 weeks | Administered 2 times 1 baseline, then 12 weeks later.
  The NPI-Q is a structured interview with a caregiver or qualified study partner (defined as having direct contact > 2 days/week) that evaluates both presence and severity of 12 neuropsychiatric features which include: delusions, hallucinations, dysphoria, anxiety, agitation/aggression, euphoria, disinhibition, irritability, lability, apathy, aberrant motor behavior, night-time behavior, and appetite/ eating changes. If the response to the domain question is "No", the informant goes to the next question. If "Yes", the informant then rates both the Severity of the symptoms present within the last month on a 3-point scale ranging from 1 to 3 (mild to severe). Change in overall NPI-Q score between baseline and at 12 weeks will be the primary outcome measure.

SECONDARY OUTCOMES:
Change from Baseline Neuropsychiatric Inventory Questionnaire subscale of caregiver distress at 12 weeks | Administered 2 times 1 baseline, then 12 weeks later.
  The NPI-Q is a structured interview with a caregiver or qualified study partner (defined as having direct contact > 2 days/week) that evaluates both presence and severity of 12 neuropsychiatric features which include: delusions, hallucinations, dysphoria, anxiety, agitation/aggression, euphoria, disinhibition, irritability, lability, apathy, aberrant motor behavior, night-time behavior, and appetite/ eating changes. A modification of the original NPI is the addition of a Caregiver Distress Scale for evaluating the psychological impact of neuropsychiatric symptoms reported to be present. For each feature the caregiver distress score ranges from 1-5 (No distress to extreme distress). The caregiver distress subscale score is the sum of the distress scores for each of the 12 features. Change in overall NPI-Q subscale of caregiver distress score which is the between baseline and at 12 weeks will be a secondary outcome measure.
Change from Baseline Zarit Burden Interview Screening Version at 12 weeks | Administered 2 times 1 baseline, then 12 weeks later.
  The Zarit Burden Interview (ZBI) Screening Version is a popular caregiver self-report measure used by many aging agencies, and originated as a 29-item questionnaire. The revised screening version contains 4 items and has been validated. Each item on the interview is a statement which the caregiver is asked to endorse using a 4-point scale. Response options range from 0 (Never) to 4 (Nearly Always). Change in overall ZBI score between baseline and at 12 weeks will be a secondary outcome measure.
Change from Baseline Short Form Health Survey 12-Item at 12 weeks | Administered 2 times 1 baseline, then 12 weeks later.
  The 12-Item Short Form Health Survey (SF-12) is a 12-item validated shortened version of the SF-36 and was designed to provide a health-related quality of life (HRQL) measure that was quick and easy to administer in large population studies. The SF-12 contains a subset of the 12 items from the SF-36 and information from this subset of questions is used to construct a physical and mental component summary score (PCS and MCS, respectively). Change in overall SF-12 score between baseline and at 12 weeks will be a secondary outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Lynne Shinto, N.D., M.P.H., Principal Investigator — Oregon Health and Science University; Sarah Goodlin, M.D., Principal Investigator — Portland VA, Oregon Health and Science University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hersch EC, Falzgraf S. Management of the behavioral and psychological symptoms of dementia. Clin Interv Aging. 2007;2(4):611-21. doi: 10.2147/cia.s1698. PMID 18225462
- [Background] de Oliveira AM, Radanovic M, de Mello PC, Buchain PC, Vizzotto AD, Celestino DL, Stella F, Piersol CV, Forlenza OV. Nonpharmacological Interventions to Reduce Behavioral and Psychological Symptoms of Dementia: A Systematic Review. Biomed Res Int. 2015;2015:218980. doi: 10.1155/2015/218980. Epub 2015 Nov 29. PMID 26693477
- [Background] Dorey JM, Beauchet O, Thomas Anterion C, Rouch I, Krolak-Salmon P, Gaucher J, Gonthier R, Akiskal HS. Behavioral and psychological symptoms of dementia and bipolar spectrum disorders: review of the evidence of a relationship and treatment implications. CNS Spectr. 2008 Sep;13(9):796-803. doi: 10.1017/s1092852900013924. PMID 18849899
- [Background] Adams BE, Tunis SL, Edell WS. Assessing antipsychotic effectiveness in dementia with the factor structure of the Psychogeriatric Dependency Rating Scale (PGDRS). J Am Med Dir Assoc. 2003 Mar-Apr;4(2):61-6. doi: 10.1097/01.JAM.0000052521.47659.7E. PMID 12807576
- [Background] Herrmann N. Recommendations for the management of behavioral and psychological symptoms of dementia. Can J Neurol Sci. 2001 Feb;28 Suppl 1:S96-107. doi: 10.1017/s0317167100001268. PMID 11237317
- [Background] Kar N. Behavioural and Psychological Symptoms of Dementia. In: Kar N, Jolley D, Misra N, editors. Handbook of Dementia. Hyderabad: Paras Medical Publisher; 2005. pp. 54-74.
- [Background] Wynn ZJ, Cummings JL. Cholinesterase inhibitor therapies and neuropsychiatric manifestations of Alzheimer's disease. Dement Geriatr Cogn Disord. 2004;17(1-2):100-8. doi: 10.1159/000074281. Epub 2003 Oct 15. PMID 14564129
- [Background] Mori T, Koyama N, Guillot-Sestier MV, Tan J, Town T. Ferulic acid is a nutraceutical beta-secretase modulator that improves behavioral impairment and alzheimer-like pathology in transgenic mice. PLoS One. 2013;8(2):e55774. doi: 10.1371/journal.pone.0055774. Epub 2013 Feb 8. PMID 23409038
- [Background] Kimura T, Hayashida H, Murata M, Takamatsu J. Effect of ferulic acid and Angelica archangelica extract on behavioral and psychological symptoms of dementia in frontotemporal lobar degeneration and dementia with Lewy bodies. Geriatr Gerontol Int. 2011 Jul;11(3):309-14. doi: 10.1111/j.1447-0594.2010.00687.x. Epub 2011 Jan 28. PMID 21272180
- [Background] Lin SY, Lewis FM. Dementia friendly, dementia capable, and dementia positive: concepts to prepare for the future. Gerontologist. 2015 Apr;55(2):237-44. doi: 10.1093/geront/gnu122. Epub 2015 Feb 15. PMID 26035599
- [Background] Lyketsos CG, Lopez O, Jones B, Fitzpatrick AL, Breitner J, DeKosky S. Prevalence of neuropsychiatric symptoms in dementia and mild cognitive impairment: results from the cardiovascular health study. JAMA. 2002 Sep 25;288(12):1475-83. doi: 10.1001/jama.288.12.1475. PMID 12243634
- [Background] Kales HC, Kim HM, Zivin K, Valenstein M, Seyfried LS, Chiang C, Cunningham F, Schneider LS, Blow FC. Risk of mortality among individual antipsychotics in patients with dementia. Am J Psychiatry. 2012 Jan;169(1):71-9. doi: 10.1176/appi.ajp.2011.11030347. Epub 2011 Oct 31. PMID 22193526
- [Background] Haupt M, Kurz A, Janner M. A 2-year follow-up of behavioural and psychological symptoms in Alzheimer's disease. Dement Geriatr Cogn Disord. 2000 May-Jun;11(3):147-52. doi: 10.1159/000017228. PMID 10765045
- [Background] Wang F, Feng TY, Yang S, Preter M, Zhou JN, Wang XP. Drug Therapy for Behavioral and Psychological Symptoms of Dementia. Curr Neuropharmacol. 2016;14(4):307-13. doi: 10.2174/1570159x14666151208114232. PMID 26644152
- [Background] Prince M, Bryce R, Albanese E, Wimo A, Ribeiro W, Ferri CP. The global prevalence of dementia: a systematic review and metaanalysis. Alzheimers Dement. 2013 Jan;9(1):63-75.e2. doi: 10.1016/j.jalz.2012.11.007. PMID 23305823
- [Background] Nielsen RE, Lolk A, M Rodrigo-Domingo, Valentin JB, Andersen K. Antipsychotic treatment effects on cardiovascular, cancer, infection, and intentional self-harm as cause of death in patients with Alzheimer's dementia. Eur Psychiatry. 2017 May;42:14-23. doi: 10.1016/j.eurpsy.2016.11.013. Epub 2016 Dec 12. PMID 28199869
- [Background] Wang PS, Schneeweiss S, Avorn J, Fischer MA, Mogun H, Solomon DH, Brookhart MA. Risk of death in elderly users of conventional vs. atypical antipsychotic medications. N Engl J Med. 2005 Dec 1;353(22):2335-41. doi: 10.1056/NEJMoa052827. PMID 16319382
- [Background] Trifiro G, Verhamme KM, Ziere G, Caputi AP, Ch Stricker BH, Sturkenboom MC. All-cause mortality associated with atypical and typical antipsychotics in demented outpatients. Pharmacoepidemiol Drug Saf. 2007 May;16(5):538-44. doi: 10.1002/pds.1334. PMID 17036366
- [Background] Sosulski, F., Krygier, K., & Hogge, L. (1982). Free, esterified, and insoluble-bound phenolic acids. 3. Composition of phenolic acids in cereal and potato flours. Journal of Agricultural and Food Chemistry, 30(2), 337-340.
- [Background] Lempereur, I., Rouau, X., & Abecassis, J. (1997). Arabinoxylan and ferulic acid variation in durum wheat (Triticum durum Desf.) grain and distribution in mill streams. J. Cereal Sci, 25, 103-110.
- [Background] Kikuzaki H, Hisamoto M, Hirose K, Akiyama K, Taniguchi H. Antioxidant properties of ferulic acid and its related compounds. J Agric Food Chem. 2002 Mar 27;50(7):2161-8. doi: 10.1021/jf011348w. PMID 11902973
- [Background] Kanski J, Aksenova M, Stoyanova A, Butterfield DA. Ferulic acid antioxidant protection against hydroxyl and peroxyl radical oxidation in synaptosomal and neuronal cell culture systems in vitro: structure-activity studies. J Nutr Biochem. 2002 May;13(5):273-281. doi: 10.1016/s0955-2863(01)00215-7. PMID 12015157
- [Background] Sgarbossa A, Giacomazza D, di Carlo M. Ferulic Acid: A Hope for Alzheimer's Disease Therapy from Plants. Nutrients. 2015 Jul 15;7(7):5764-82. doi: 10.3390/nu7075246. PMID 26184304
- [Background] Srinivasan M, Sudheer AR, Menon VP. Ferulic Acid: therapeutic potential through its antioxidant property. J Clin Biochem Nutr. 2007 Mar;40(2):92-100. doi: 10.3164/jcbn.40.92. PMID 18188410
- [Background] Ou L, Kong LY, Zhang XM, Niwa M. Oxidation of ferulic acid by Momordica charantia peroxidase and related anti-inflammation activity changes. Biol Pharm Bull. 2003 Nov;26(11):1511-6. doi: 10.1248/bpb.26.1511. PMID 14600392
- [Background] He XX, Yang XH, Ou RY, Ouyang Y, Wang SN, Chen ZW, Wen SJ, Pi RB. Synthesis and evaluation of multifunctional ferulic and caffeic acid dimers for Alzheimer's disease. Nat Prod Res. 2017 Mar;31(6):734-737. doi: 10.1080/14786419.2016.1219862. Epub 2016 Aug 17. PMID 27531418
- [Background] Singh JC, Kakalij RM, Kshirsagar RP, Kumar BH, Komakula SS, Diwan PV. Cognitive effects of vanillic acid against streptozotocin-induced neurodegeneration in mice. Pharm Biol. 2015 May;53(5):630-6. doi: 10.3109/13880209.2014.935866. Epub 2014 Dec 4. PMID 25472801
- [Background] Jacobson, E. A., Newmark, H., Baptista, J., & Bruce, W. R. (1983). A preliminary investigation of the metabolism of dietary phenolics in humans [Urinary metabolites of caffeic and ferulic acid]. Nutrition Reports International.
- [Background] Sadigh-Eteghad S, Sabermarouf B, Majdi A, Talebi M, Farhoudi M, Mahmoudi J. Amyloid-beta: a crucial factor in Alzheimer's disease. Med Princ Pract. 2015;24(1):1-10. doi: 10.1159/000369101. Epub 2014 Nov 27. PMID 25471398
- [Background] Tan RH, Kril JJ, Yang Y, Tom N, Hodges JR, Villemagne VL, Rowe CC, Leyton CE, Kwok JBJ, Ittner LM, Halliday GM. Assessment of amyloid beta in pathologically confirmed frontotemporal dementia syndromes. Alzheimers Dement (Amst). 2017 May 29;9:10-20. doi: 10.1016/j.dadm.2017.05.005. eCollection 2017. PMID 28653036
- [Background] Simic G, Babic Leko M, Wray S, Harrington C, Delalle I, Jovanov-Milosevic N, Bazadona D, Buee L, de Silva R, Di Giovanni G, Wischik C, Hof PR. Tau Protein Hyperphosphorylation and Aggregation in Alzheimer's Disease and Other Tauopathies, and Possible Neuroprotective Strategies. Biomolecules. 2016 Jan 6;6(1):6. doi: 10.3390/biom6010006. PMID 26751493
- [Background] Porat Y, Abramowitz A, Gazit E. Inhibition of amyloid fibril formation by polyphenols: structural similarity and aromatic interactions as a common inhibition mechanism. Chem Biol Drug Des. 2006 Jan;67(1):27-37. doi: 10.1111/j.1747-0285.2005.00318.x. PMID 16492146
- [Background] Ono K, Hirohata M, Yamada M. Ferulic acid destabilizes preformed beta-amyloid fibrils in vitro. Biochem Biophys Res Commun. 2005 Oct 21;336(2):444-9. doi: 10.1016/j.bbrc.2005.08.148. PMID 16153607
- [Background] Sul D, Kim HS, Lee D, Joo SS, Hwang KW, Park SY. Protective effect of caffeic acid against beta-amyloid-induced neurotoxicity by the inhibition of calcium influx and tau phosphorylation. Life Sci. 2009 Feb 27;84(9-10):257-62. doi: 10.1016/j.lfs.2008.12.001. Epub 2008 Dec 7. PMID 19101570
- [Background] Ou, S., & Kwok, K. C. (2004). Ferulic acid: pharmaceutical functions, preparation and applications in foods. Journal of the Science of Food and Agriculture, 84(11), 1261-1269.
- [Background] Bartus RT, Dean RL 3rd, Beer B, Lippa AS. The cholinergic hypothesis of geriatric memory dysfunction. Science. 1982 Jul 30;217(4558):408-14. doi: 10.1126/science.7046051.
- [Background] Bartolini M, Bertucci C, Cavrini V, Andrisano V. beta-Amyloid aggregation induced by human acetylcholinesterase: inhibition studies. Biochem Pharmacol. 2003 Feb 1;65(3):407-16. doi: 10.1016/s0006-2952(02)01514-9. PMID 12527333
- [Background] Alvarez A, Opazo C, Alarcon R, Garrido J, Inestrosa NC. Acetylcholinesterase promotes the aggregation of amyloid-beta-peptide fragments by forming a complex with the growing fibrils. J Mol Biol. 1997 Sep 26;272(3):348-61. doi: 10.1006/jmbi.1997.1245. PMID 9325095
- [Background] Bao F, Wicklund L, Lacor PN, Klein WL, Nordberg A, Marutle A. Different beta-amyloid oligomer assemblies in Alzheimer brains correlate with age of disease onset and impaired cholinergic activity. Neurobiol Aging. 2012 Apr;33(4):825.e1-13. doi: 10.1016/j.neurobiolaging.2011.05.003. Epub 2011 Jun 17. PMID 21683475
- [Background] Wszelaki N, Paradowska K, Jamroz MK, Granica S, Kiss AK. Bioactivity-guided fractionation for the butyrylcholinesterase inhibitory activity of furanocoumarins from Angelica archangelica L. roots and fruits. J Agric Food Chem. 2011 Sep 14;59(17):9186-93. doi: 10.1021/jf201971s. Epub 2011 Aug 9. PMID 21786787
- [Background] Sigurdsson S, Gudbjarnason S. Effect of oral imperatorin on memory in mice. Biochem Biophys Res Commun. 2013 Nov 15;441(2):318-20. doi: 10.1016/j.bbrc.2013.10.036. Epub 2013 Oct 16. PMID 24140410
- [Background] Budzynska B, Boguszewska-Czubara A, Kruk-Slomka M, Skalicka-Wozniak K, Michalak A, Musik I, Biala G, Glowniak K. Effects of imperatorin on nicotine-induced anxiety- and memory-related responses and oxidative stress in mice. Physiol Behav. 2013 Oct 2;122:46-55. doi: 10.1016/j.physbeh.2013.08.019. Epub 2013 Aug 30. PMID 23999469
- [Background] Sigurdsson S, Geirsson G, Gudmundsdottir H, Egilsdottir PB, Gudbjarnason S. A parallel, randomized, double-blind, placebo-controlled study to investigate the effect of SagaPro on nocturia in men. Scand J Urol. 2013 Feb;47(1):26-32. doi: 10.3109/00365599.2012.695390. Epub 2012 Jul 2. PMID 23323790
- [Background] Kanaya, K. (2010). Effects of ferulic acid and Angelica archangelica extract (Feruguard) in patients with Alzheimer's disease. Alzheimer's & Dementia: The Journal of the Alzheimer's Association, 6(4), S548.
- [Background] Kimura, T. (2014). A Pilot Study of Tretment with Ferulic Acid and Angelica archangelica Extract for Cognitive Impairment. Journal of New Remedies & Clinics, 63(11), 1848-1855.
- [Background] Cummings JL, Mega M, Gray K, Rosenberg-Thompson S, Carusi DA, Gornbein J. The Neuropsychiatric Inventory: comprehensive assessment of psychopathology in dementia. Neurology. 1994 Dec;44(12):2308-14. doi: 10.1212/wnl.44.12.2308. PMID 7991117
- [Background] Kaufer DI, Cummings JL, Ketchel P, Smith V, MacMillan A, Shelley T, Lopez OL, DeKosky ST. Validation of the NPI-Q, a brief clinical form of the Neuropsychiatric Inventory. J Neuropsychiatry Clin Neurosci. 2000 Spring;12(2):233-9. doi: 10.1176/jnp.12.2.233. PMID 11001602
- [Background] Morris JC. The Clinical Dementia Rating (CDR): current version and scoring rules. Neurology. 1993 Nov;43(11):2412-4. doi: 10.1212/wnl.43.11.2412-a. No abstract available. PMID 8232972
- [Background] Salthouse TA. What do adult age differences in the Digit Symbol Substitution Test reflect? J Gerontol. 1992 May;47(3):P121-8. doi: 10.1093/geronj/47.3.p121. PMID 1573192
- [Background] Smith T, Gildeh N, Holmes C. The Montreal Cognitive Assessment: validity and utility in a memory clinic setting. Can J Psychiatry. 2007 May;52(5):329-32. doi: 10.1177/070674370705200508. PMID 17542384
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Gandek B, Ware JE, Aaronson NK, Apolone G, Bjorner JB, Brazier JE, Bullinger M, Kaasa S, Leplege A, Prieto L, Sullivan M. Cross-validation of item selection and scoring for the SF-12 Health Survey in nine countries: results from the IQOLA Project. International Quality of Life Assessment. J Clin Epidemiol. 1998 Nov;51(11):1171-8. doi: 10.1016/s0895-4356(98)00109-7. PMID 9817135
- [Background] Zarit SH, Reever KE, Bach-Peterson J. Relatives of the impaired elderly: correlates of feelings of burden. Gerontologist. 1980 Dec;20(6):649-55. doi: 10.1093/geront/20.6.649. No abstract available. PMID 7203086
- [Background] Bedard M, Molloy DW, Squire L, Dubois S, Lever JA, O'Donnell M. The Zarit Burden Interview: a new short version and screening version. Gerontologist. 2001 Oct;41(5):652-7. doi: 10.1093/geront/41.5.652. PMID 11574710
- [Background] National Cancer Institute (NCI). Dietary Screener Questionnaire (DSQ) website:<http://riskfactor.cancer.gov/studies/nhanes/dietscreen/questionnaires.html>. Accessed 6 February 2012.
- [Background] Kivipelto M, Helkala EL, Laakso MP, Hanninen T, Hallikainen M, Alhainen K, Iivonen S, Mannermaa A, Tuomilehto J, Nissinen A, Soininen H. Apolipoprotein E epsilon4 allele, elevated midlife total cholesterol level, and high midlife systolic blood pressure are independent risk factors for late-life Alzheimer disease. Ann Intern Med. 2002 Aug 6;137(3):149-55. doi: 10.7326/0003-4819-137-3-200208060-00006. PMID 12160362
- [Background] Tan ZS, Seshadri S, Beiser A, Wilson PW, Kiel DP, Tocco M, D'Agostino RB, Wolf PA. Plasma total cholesterol level as a risk factor for Alzheimer disease: the Framingham Study. Arch Intern Med. 2003 May 12;163(9):1053-7. doi: 10.1001/archinte.163.9.1053. PMID 12742802
- [Background] Gibson Wood W, Eckert GP, Igbavboa U, Muller WE. Amyloid beta-protein interactions with membranes and cholesterol: causes or casualties of Alzheimer's disease. Biochim Biophys Acta. 2003 Mar 10;1610(2):281-90. doi: 10.1016/s0005-2736(03)00025-7. PMID 12648781
- [Background] Hixson JE, Vernier DT. Restriction isotyping of human apolipoprotein E by gene amplification and cleavage with HhaI. J Lipid Res. 1990 Mar;31(3):545-8. PMID 2341813